CLINICAL TRIAL: NCT01305720
Title: The Effect of Mydriatic Eye Drops on Cerebral and Mesenteric Oxygenation in Preterm Infants
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zekai Tahir Burak Women's Health Research and Education Hospital (Other)
Responsible Party: Zekai Tahir Burak Maternity and Teaching Hospital, Zekai Tahir Burak Maternity and Teaching Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 734
Record Dates: First submitted 2011-02-28; First posted 2011-03-01 (Estimated); Last update posted 2011-03-01 (Estimated); Status verified 2011-02

CONDITIONS: Prematurity of Fetus
Keywords: mydriatic; NIRS; preterm; eye drops; cerebral; mesenteric oxygenation
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: near infrared spectroscopy: invos 5100 — NIRS device used in this study, the optical field includes a volume of tissue approximately 2 cm deep to the surface probe with a 4-mm source-detector distance, and thus, organ-specific monitoring is feasible in small patients. With informed consent, the investigators applied NIRS probes to the forehead and abdomen for cerebral (rSO2C) and abdominal (rSO2P) regional oxygen saturation measurements.

SUMMARY:
Near infrared spectroscopy offers the possibility of noninvasive and continuous bedside investigation of cerebral and mesenteric oxygenation in newborn infants. Using this technique the investigators investigated the effect of mydriatic eye drops on cerebral and mesenteric oxygenation in preterm infants

DETAILED DESCRIPTION:
The cerebral and mesenteric oxygenation will be measured by NIRS before, during and after the mydriatic eye drops are instilled.

ELIGIBILITY:
Inclusion Criteria:

1. < 32 gestational age and/or < 1500gr.
2. ≥ 28th day preterm infants
3. Instilled mydriatic eye drops for ROP examination

Exclusion Criteria:

1. Sepsis
2. Shock
3. Severe intracranial hemorrhage
4. NEC
5. Abdominal and cranial surgery

Ages: 28 Days to 90 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2011-03; Primary Completion 2011-06 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
The Effect of Mydriatic Eye Drops on Cerebral and mesenteric Oxygenation | one year
  By NIRS cerebral and mesenteric oxygenation will be measured before, during and after mydriatic eye drops are instilled.

CONTACTS AND LOCATIONS:
Locations (1):
- Zekai Tahir Burak Maternity and Teaching Hospital, Ankara, Turkey (Türkiye)